CLINICAL TRIAL: NCT01519674
Title: A 24 Week Randomised, Open Label, 3 Parallel-group Comparison of Once and Twice Daily Biphasic Insulin Aspart (BIAsp) 30 Plus Sitagliptin and Twice Daily BIAsp 30, All in Combination With Metformin in Insulin naïve Type 2 Diabetic Subjects Inadequately Controlled on Sitagliptin and Metformin
Brief Title: Treatment Intensification With Biphasic Insulin Aspart 30 in Subjects With Type 2 Diabetes Inadequately Controlled on Sitagliptin and Metformin
Acronym: SIT2MIX
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BIASP-3963; U1111-1125-0850 (Other: WHO); 2011-004930-33 (EudraCT Number)
Record Dates: First submitted 2012-01-24; First posted 2012-01-27 (Estimated); Results first posted 2014-11-10 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — insulin aspart, insulin aspart protamine drug combination 30:70; Sitagliptin Phosphate; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- BIAsp 30 BID + sitagliptin + metformin (Active Comparator)
  Interventions: Drug: biphasic insulin aspart 30; Drug: sitagliptin; Drug: metformin
- BIAsp 30 BID + metformin (Active Comparator)
  Interventions: Drug: biphasic insulin aspart 30; Drug: metformin
- BIAsp 30 OD + sitagliptin + metformin (Active Comparator)
  Interventions: Drug: biphasic insulin aspart 30; Drug: sitagliptin; Drug: metformin

INTERVENTIONS:
Drug: biphasic insulin aspart 30 — BIAsp 30 will be injected subcutaneously (under the skin) twice daily. Individually adjusted dose.
  Arms: BIAsp 30 BID + metformin; BIAsp 30 BID + sitagliptin + metformin
Drug: biphasic insulin aspart 30 — BIAsp 30 will be injected subcutaneously (under the skin) once daily. Individually adjusted dose.
  Arms: BIAsp 30 OD + sitagliptin + metformin
Drug: sitagliptin — Subjects will continue on their pre-trial sitagliptin treatment.
  Arms: BIAsp 30 BID + sitagliptin + metformin; BIAsp 30 OD + sitagliptin + metformin
Drug: metformin — Subjects will continue on their pre-trial metformin treatment.

SUMMARY:
This trial is conducted in Asia, Europe, Oceania and South America. The aim of this clinical trial is to generate data demonstrating how to intensify diabetes treatment using BIAsp 30 (biphasic insulin aspart 30) by adding or substituting BIAsp 30 to sitagliptin in various regimens for type 2 patients inadequately controlled on sitagliptin and metformin (with or without other oral anti-diabetic drugs (OADs)).

The trial is conducted as a phase 4 trial in the majority of the participating countries. However, in some countries the trial is conducted as phase 3b.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with type 2 diabetes for a minimum of 6 months prior to screening (Visit 1)
* Stable treatment with a total daily dose of at least 1000 mg of metformin (with or without additional oral anti-diabetic drugs (OADs) treatment). The metformin dose must have been unchanged for at least 3 months prior to screening (Visit 1)
* Stable treatment with a total daily dose of at least 100 mg sitagliptin. The sitagliptin dose must have been unchanged for at least 3 months prior to screening (Visit 1)
* Subject is insulin-naïve (never previously treated with insulin). (However, short term insulin use due to intermittent illness of up to 14 days or insulin treatment for gestational diabetes is allowed)
* HbA1c (glycosylated haemoglobin) between 7.0 to 10.0 % (53-86 mmol/mol) (both inclusive) by central laboratory analysis demonstrating inadequate control on sitagliptin and metformin (with or without other OADs)
* Body Mass Index (BMI) below or equal to 40.0 kg/m^2
* Able and willing to eat at least 2 meals (breakfast and dinner) every day during the trial

Exclusion Criteria:

* Treatment with thiazolidinedione (TZD) or glucagon-like-peptide-1 (GLP-1) receptor agonist within the last 3 months prior to screening (Visit 1)
* Cardiac disease within the last 6 months prior to screening (Visit 1), defined as: decompensated heart failure New York Heart Association (NYHA) class III or IV; unstable angina pectoris; or myocardial infarction
* Severe hypertension, systolic blood pressure equal to or above 180 mm Hg or diastolic blood pressure equal to or above 100 mm Hg, after 5 minutes rest in the sitting position using mean value of 3 measurements at screening (Visit 1)
* Anticipated change of dose of any systemic treatment with products, which in the trial physician's opinion could interfere with glucose metabolism (e.g., systemic corticosteroids)
* Clinically significant diseases (except for conditions associated with type 2 diabetes) which, in the trial physician's opinion may confound the results of the trial or pose additional risk in administering trial product(s)
* Impaired hepatic function as indicated by aspartate aminotransferase (ASAT) or alanine aminotransferase (ALAT) above 2.5 times the upper normal range, according to central laboratory reference ranges
* Impaired renal function as indicated by serum creatinine levels equal to or above 133 micromol/L (1.5 mg/dL) for males and equal to or above 124 micromol/L (1.4 mg/dL) for females or estimated creatinine clearance below 60 mL/min, based on the Cockroft & Gault formula and according to local practise for metformin use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 582 (Actual)
Dates: Start 2012-06; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (48):
- Argentina (4):
  - Novo Nordisk Investigational Site, Buenos Aires
  - Novo Nordisk Investigational Site, Caba
  - Novo Nordisk Investigational Site, Mar del Plata
  - Novo Nordisk Investigational Site, Morón
- Australia (2):
  - Novo Nordisk Investigational Site, Broadmeadow, New South Wales
  - Novo Nordisk Investigational Site, Coffs Harbour, New South Wales
- Brazil (5):
  - Novo Nordisk Investigational Site, São Paulo, São Paulo
  - Novo Nordisk Investigational Site, Brasília
  - Novo Nordisk Investigational Site, Curitiba
  - Novo Nordisk Investigational Site, Fortaleza
  - Novo Nordisk Investigational Site, Porto Alegre
- Greece (3):
  - Novo Nordisk Investigational Site, Alexandroupoli
  - Novo Nordisk Investigational Site, Athens
  - Novo Nordisk Investigational Site, Thessaloniki
- India (16):
  - Novo Nordisk Investigational Site, Hyderabad, Andhra Pradesh
  - Novo Nordisk Investigational Site, Visakhapatnam, Andhra Pradesh
  - Novo Nordisk Investigational Site, Ahmedabad, Gujarat
  - Novo Nordisk Investigational Site, Bangalore, Karnataka
  - Novo Nordisk Investigational Site, Calicut, Kerala
  - Novo Nordisk Investigational Site, Trivandrum, Kerala
  - Novo Nordisk Investigational Site, Nagpur, Maharashtra
  - Novo Nordisk Investigational Site, New Delhi, New Delhi
  - Novo Nordisk Investigational Site, Amritsar, Punjab
  - Novo Nordisk Investigational Site, Chennai, Tamil Nadu
  - Novo Nordisk Investigational Site, Coimbatore, Tamil Nadu
  - Novo Nordisk Investigational Site, Trichy, Tamil Nadu
  - Novo Nordisk Investigational Site, Kanpur, Uttar Pradesh
  - Novo Nordisk Investigational Site, Noida, Uttar Pradesh
  - Novo Nordisk Investigational Site, Varanasi, Uttar Pradesh
  - Novo Nordisk Investigational Site, Kolkata, West Bengal
- Malaysia (2):
  - Novo Nordisk Investigational Site, George Town
  - Novo Nordisk Investigational Site, Seremban
- Portugal (4):
  - Novo Nordisk Investigational Site, Coimbra
  - Novo Nordisk Investigational Site, Lisbon
  - Novo Nordisk Investigational Site, Matosinhos Municipality
  - Novo Nordisk Investigational Site, Porto
- South Korea (7):
  - Novo Nordisk Investigational Site, Goyang
  - Novo Nordisk Investigational Site, Jeonju
  - Novo Nordisk Investigational Site, Pusan
  - Novo Nordisk Investigational Site, Pyungchon-Dong 896, Dongan-Gu
  - Novo Nordisk Investigational Site, Seoul
  - Novo Nordisk Investigational Site, Suwon
  - Novo Nordisk Investigational Site, Ulsan
- Thailand (3):
  - Novo Nordisk Investigational Site, Bangkok
  - Novo Nordisk Investigational Site, Chiang Mai
  - Novo Nordisk Investigational Site, Khon Kaen
- Turkey (Türkiye) (2):
  - Novo Nordisk Investigational Site, Antalya
  - Novo Nordisk Investigational Site, Istanbul

REFERENCES:
- [Result] Linjawi S, Sothiratnam R, Sari R, Andersen H, Hiort LC, Rao P. The study of once- and twice-daily biphasic insulin aspart 30 (BIAsp 30) with sitagliptin, and twice-daily BIAsp 30 without sitagliptin, in patients with type 2 diabetes uncontrolled on sitagliptin and metformin-The Sit2Mix trial. Prim Care Diabetes. 2015 Oct;9(5):370-6. doi: 10.1016/j.pcd.2014.11.001. Epub 2014 Dec 3. PMID 25488587
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 60 sites in 10 countries as follows:
  Argentina (6); Australia (2); Brazil (4); Greece (5); India (17); Malaysia (3); Portugal (6); Republic of Korea (7); Thailand (5); Turkey (5)
Pre-assignment Details: Subjects on pre-trial metformin (1000 mg/day) (± additional OAD treatment) continued their medication. Subjects on pre-trial sitagliptin (100 mg/day) either continued or discontinued their sitagliptin treatment depending on the treatment group the subjects were randomised to.
Groups:
- BID + Met: Biphasic insulin aspart 30 (BIAsp 30) was injected twice daily, 6 U before breakfast and 6 U before dinner (evening meal), subcutaneously (under the skin) for 24 weeks. Dosing of BIAsp 30 was adjusted individually according to the titration guideline and the subject's self-measured plasma glucose (SMPG) levels. Subjects continued on their pre-trial metformin (1000 mg/day) treatment.
- BID + Sita + Met: Biphasic insulin aspart 30 (BIAsp 30) was injected twice daily, 6 U before breakfast and 6 U before dinner (evening meal), subcutaneously (under the skin) for 24 weeks. Dosing of BIAsp 30 was adjusted individually according to the titration guideline and the subject's self-measured plasma glucose (SMPG) levels. Subjects continued on their pre-trial metformin (1000 mg/day) and sitagliptin (100 mg/day) treatments.
- OD + Sita + Met: Biphasic insulin aspart 30 (BIAsp 30) was injected once daily, 12 U before dinner (evening meal), subcutaneously (under the skin) for 24 weeks. Dosing of BIAsp 30 was adjusted individually according to the titration guideline and the subject's self-measured plasma glucose (SMPG) levels. Subjects continued on their pre-trial metformin (1000 mg/day) and sitagliptin (100 mg/day) treatments.
Period: Overall Study
Arm/Group | BID + Met | BID + Sita + Met | OD + Sita + Met
Started | 194 | 195 | 193
Exposed | 192 | 193 | 190
Completed | 173 | 182 | 181
Not Completed | 21 | 13 | 12
Not completed — Adverse Event | 3 | 3 | 0
Not completed — Lack of Efficacy | 1 | 1 | 1
Not completed — Protocol Violation | 0 | 3 | 1
Not completed — Withdrawal Criteria | 7 | 2 | 7
Not completed — Unsclassified | 10 | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BID + Met | BID + Sita + Met | OD + Sita + Met | Total
Number analyzed (Participants) | 194 | 195 | 193 | 582
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.8 (9.5) | 56.3 (10.2) | 55.7 (10.4) | 55.6 (10.0)
Gender [Count of Participants; unit: Participants]
  Female | 83 | 101 | 97 | 281
  Male | 111 | 94 | 96 | 301
Body Weight [Mean (Standard Deviation); unit: kg] | 79.4 (15.8) | 78.3 (16.1) | 77.5 (16.8) | 78.4 (16.2)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 29.3 (4.3) | 29.4 (4.5) | 29.4 (5.0) | 29.4 (4.6)
Glycosylated haemoglobin (HbA1c) [Mean (Standard Deviation); unit: Percent (%) glycosylated haemoglobin] | 8.4 (0.8) | 8.4 (0.8) | 8.4 (0.8) | 8.4 (0.8)
Fasting plasma glucose (FPG) [Mean (Standard Deviation); unit: mmol/L] | 8.9 (2.2) | 9.3 (2.8) | 8.7 (2.7) | 9.0 (2.6)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in HbA1c (Glycosylated Haemoglobin)
Description: Estimated mean change from baseline in HbA1c after 24 weeks of treatment.
Time Frame: Week 0 to Week 24
Population: Full analysis set (FAS) included all randomised subjects and missing data were imputed using last observation carried forward (LOCF). 559 subjects contributed to the statistical analysis at Week 24.
Measure: Least Squares Mean (Standard Error); unit: percentage of glycosylated haemoglobin
Arm/Group | BID + Met | BID + Sita + Met | OD + Sita + Met
Number analyzed (Participants) | 183 | 189 | 187
percentage of glycosylated haemoglobin | -1.27 (0.07) | -1.51 (0.07) | -1.15 (0.07)
Statistical Analysis 1: Comparison: BID + Met vs BID + Sita + Met; The null-hypothesis (H0) was tested against the alternative hypothesis (HA) in each of the comparisons as given by: H0: D = 0% against HA: D ≠ 0% D being the mean treatment difference for change from baseline in HbA1c after 24 weeks of treatment between the two treatment group comparisons (BID+Met and BID+Sita+Met); Test type: Superiority or Other; p = 0.011, Regression, Linear — No corrections for multiplicity were performed; Estimated treatment difference = 0.24, 95% CI [0.06 to 0.43]
Statistical Analysis 2: Comparison: BID + Met vs OD + Sita + Met; The null-hypothesis (H0) was tested against the alternative hypothesis (HA) in each of the comparisons as given by: H0: D = 0% against HA: D ≠ 0% D being the mean treatment difference for change from baseline in HbA1c after 24 weeks of treatment between the two treatment group comparisons (BID+Sita+Met and OD+Sita+Met); Test type: Superiority or Other; p = 0.231, Regression, Linear; Estimated treatment difference = -0.11, 95% CI [-0.30 to 0.07]
Statistical Analysis 3: Comparison: BID + Sita + Met vs OD + Sita + Met; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.001, Regression, Linear; Estimated treatment difference = -0.36, 95% CI [-0.54 to -0.17]

2. Secondary Outcome: Responder for HbA1c, Proportion of Subjects Achieving Pre-defined HbA1c Targets (HbA1c < 7.0%)
Description: Proportion of subjects achieving HbA1c below 7.0% after 24 weeks of treatment
Time Frame: After 24 weeks of treatment
Population: as for outcome 1
Measure: Number; unit: percentage (%) of subjects
Arm/Group | BID + Met | BID + Sita + Met | OD + Sita + Met
Number analyzed (Participants) | 183 | 189 | 187
percentage (%) of subjects | 49.7 | 59.8 | 46.5
Statistical Analysis 1: Comparison: BID + Met vs BID + Sita + Met; Test type: Superiority or Other; p = 0.022, Regression, Logistic; Odds Ratio (OR) = 0.60, 95% CI [0.39 to 0.93]
Statistical Analysis 2: Comparison: BID + Met vs OD + Sita + Met; Test type: Superiority or Other; p = 0.618, Regression, Logistic; Odds Ratio (OR) = 1.12, 95% CI [0.73 to 1.71]
Statistical Analysis 3: Comparison: BID + Sita + Met vs OD + Sita + Met; Test type: Superiority or Other; p = 0.005, Regression, Logistic; Odds Ratio (OR) = 1.85, 95% CI [1.20 to 2.85]

3. Secondary Outcome: Responder for HbA1c, Proportion of Subjects Achieving Pre-defined HbA1c Targets (HbA1c ≤ 6.5%)
Description: Proportion of subjects achieving HbA1c equal to or below 6.5% after 24 weeks of treatment.
Time Frame: After 24 weeks of treatment
Population: as for outcome 1
Measure: Number; unit: percentage (%) of subjects
Arm/Group | BID + Met | BID + Sita + Met | OD + Sita + Met
Number analyzed (Participants) | 183 | 189 | 187
percentage (%) of subjects | 30.6 | 40.7 | 25.1
Statistical Analysis 1: Comparison: BID + Met vs BID + Sita + Met; Test type: Superiority or Other; p = 0.020, Regression, Logistic; Odds Ratio (OR) = 0.59, 95% CI [0.38 to 0.92]
Statistical Analysis 2: Comparison: BID + Met vs OD + Sita + Met; Test type: Superiority or Other; p = 0.286, Regression, Logistic; Odds Ratio (OR) = 1.29, 95% CI [0.81 to 2.07]
Statistical Analysis 3: Comparison: BID + Sita + Met vs OD + Sita + Met; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 2.20, 95% CI [1.39 to 3.47]

4. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG)
Description: Estimated mean change from baseline in fasting plasma glucose (FPG)
Time Frame: Week 0 to Week 24
Population: Full analysis set (FAS) included all randomised subjects and missing data were imputed using last observation carried forward (LOCF). 556 subjects contributed to the statistical analysis at Week 24.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | BID + Met | BID + Sita + Met | OD + Sita + Met
Number analyzed (Participants) | 181 | 188 | 187
mmol/L | -1.90 (0.14) | -2.03 (0.14) | -1.96 (0.14)
Statistical Analysis 1: Comparison: BID + Met vs BID + Sita + Met; Test type: Superiority or Other; p = 0.520, Regression, Linear; Estimated treatment difference = 0.13, 95% CI [-0.26 to 0.52]
Statistical Analysis 2: Comparison: BID + Met vs OD + Sita + Met; Test type: Superiority or Other; p = 0.788, Regression, Linear; Estimated treatment difference = 0.05, 95% CI [-0.34 to 0.45]
Statistical Analysis 3: Comparison: BID + Sita + Met vs OD + Sita + Met; Test type: Superiority or Other; p = 0.708, Regression, Linear; Estimated treatment difference = -0.07, 95% CI [-0.46 to 0.31]

5. Secondary Outcome: Prandial Plasma Glucose (PPG) Increments at Breakfast
Description: Estimated mean post prandial increments at breakfast after 24 weeks of treatment.
Time Frame: After 24 weeks of treatment
Population: Full analysis set (FAS) included all randomised subjects and missing data were imputed using last observation carried forward (LOCF). 555 subjects contributed to the statistical analysis at Week 24.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | BID + Met | BID + Sita + Met | OD + Sita + Met
Number analyzed (Participants) | 184 | 187 | 184
mmol/L | 2.01 (0.19) | 1.73 (0.19) | 2.89 (0.19)
Statistical Analysis 1: Comparison: BID + Met vs BID + Sita + Met; Test type: Superiority or Other; p = 0.291, Regression, Linear; Estimated treatment difference = 0.28, 95% CI [-0.24 to 0.81]
Statistical Analysis 2: Comparison: BID + Met vs OD + Sita + Met; Test type: Superiority or Other; p = 0.001, Regression, Linear; Estimated treatment difference = -0.88, 95% CI [-1.41 to -0.35]
Statistical Analysis 3: Comparison: BID + Sita + Met vs OD + Sita + Met; Test type: Superiority or Other; p < 0.001, Regression, Linear; Estimated treatment difference = -1.16, 95% CI [-1.69 to -0.64]

6. Secondary Outcome: Prandial Plasma Glucose (PPG) Increments at Lunch.
Description: Estimated mean post prandial increments at lunch after 24 weeks of treatment.
Time Frame: After 24 weeks of treatment
Population: Full analysis set (FAS) included all randomised subjects and missing data were imputed using last observation carried forward (LOCF). 548 subjects contributed to the statistical analysis at Week 24.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | BID + Met | BID + Sita + Met | OD + Sita + Met
Number analyzed (Participants) | 180 | 186 | 182
mmol/L | 3.05 (0.22) | 2.19 (0.21) | 2.52 (0.21)
Statistical Analysis 1: Comparison: BID + Met vs BID + Sita + Met; Test type: Superiority or Other; p = 0.005, Regression, Linear; Estimated treatment difference = 0.85, 95% CI [0.26 to 1.45]
Statistical Analysis 2: Comparison: BID + Met vs OD + Sita + Met; Test type: Superiority or Other; p = 0.085, Regression, Linear; Estimated treatment difference = 0.52, 95% CI [-0.07 to 1.12]
Statistical Analysis 3: Comparison: BID + Sita + Met vs OD + Sita + Met; Test type: Superiority or Other; p = 0.275, Regression, Linear; Estimated treatment difference = -0.33, 95% CI [-0.92 to 0.26]

7. Secondary Outcome: Prandial Plasma Glucose (PPG) Increments at Dinner.
Description: Estimated mean post prandial increments at dinner after 24 weeks of treatment.
Time Frame: After 24 weeks of treatment
Population: Full analysis set (FAS) included all randomised subjects and missing data were imputed using last observation carried forward (LOCF). 550 subjects contributed to the statistical analysis at Week 24.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | BID + Met | BID + Sita + Met | OD + Sita + Met
Number analyzed (Participants) | 178 | 188 | 184
mmol/L | 0.89 (0.21) | 1.01 (0.20) | 0.17 (0.21)
Statistical Analysis 1: Comparison: BID + Met vs BID + Sita + Met; Test type: Superiority or Other; p = 0.674, Regression, Linear; Estimated treatment difference = -0.12, 95% CI [-0.70 to 0.45]
Statistical Analysis 2: Comparison: BID + Met vs OD + Sita + Met; Test type: Superiority or Other; p = 0.015, Regression, Linear; Estimated treatment difference = 0.72, 95% CI [0.14 to 1.30]
Statistical Analysis 3: Comparison: BID + Sita + Met vs OD + Sita + Met; Test type: Superiority or Other; p = 0.004, Regression, Linear; Estimated treatment difference = 0.84, 95% CI [0.27 to 1.41]

8. Secondary Outcome: Prandial Plasma Glucose (PPG) Overall Mean Increment.
Description: Estimated overall mean post prandial increment after 24 weeks of treatment.
Time Frame: After 24 weeks of treatment
Population: Full analysis set (FAS) included all randomised subjects and missing data were imputed using last observation carried forward (LOCF). 557 subjects contributed to the statistical analysis at Week 24.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | BID + Met | BID + Sita + Met | OD + Sita + Met
Number analyzed (Participants) | 184 | 188 | 185
mmol/L | 1.97 (0.12) | 1.66 (0.12) | 1.88 (0.12)
Statistical Analysis 1: Comparison: BID + Met vs BID + Sita + Met; Test type: Superiority or Other; p = 0.080, Regression, Linear; Estimated treatment difference = 0.31, 95% CI [-0.04 to 0.65]
Statistical Analysis 2: Comparison: BID + Met vs OD + Sita + Met; Test type: Superiority or Other; p = 0.613, Regression, Linear; Estimated treatment difference = 0.09, 95% CI [-0.26 to 0.43]
Statistical Analysis 3: Comparison: BID + Sita + Met vs OD + Sita + Met; Test type: Superiority or Other; p = 0.213, Regression, Linear; Estimated treatment difference = -0.22, 95% CI [-0.56 to 0.13]

9. Secondary Outcome: Adverse Events (AEs)
Description: Rate of AEs per 100 years of patient exposure. An adverse event was defined as treatment emergent if the event had onset date on or after the first day of exposure to randomised treatment and no later than the last day of randomised treatment.
Time Frame: Week 0 to Week 24
Population: Safety analysis set included all subjects receiving at least one dose of the investigational product.
Measure: Number; unit: Events/100 years of patient exposure
Arm/Group | BID + Met | BID + Sita + Met | OD + Sita + Met
Number analyzed (Participants) | 192 | 193 | 190
Events/100 years of patient exposure
  All treatment emergent adverse events | 262.2 | 209.9 | 281.2
  Serious adverse events | 8.4 | 5.8 | 10.5
  Severe adverse events | 6.0 | 10.5 | 7.0
  Moderate adverse events | 71.0 | 74.6 | 79.7
  Mild adverse events | 185.2 | 124.8 | 194.5
  Fatal adverse events | 0 | 0 | 0

10. Secondary Outcome: Number of Treatment Emergent Hypoglycaemic Episodes (Nocturnal and Day-time) Classified Both According to the American Diabetes Association (ADA) Definition and to an Additional Definition for Minor Episodes.
Description: Number of treatment emergent hypoglycaemic episodes. Treatment emergent hypoglycaemic episode: if the onset of the episode was on or after the first day of exposure to randomised treatment and no later than the last day of randomised treatment. Nocturnal: Time of onset between 00:01 and 05:59 a.m. (both included). Additional minor hypoglycaemic episode: symptomatic or asymptomatic hypoglycaemia with blood glucose (BG) values < 2.8 mmol/L (50 mg/dL) or plasma glucose (PG) < 3.1 mmol/L (56 mg/dL), and which was handled by the subject him/herself.
Time Frame: Week 0 to Week 24
Population: Safety analysis set included all subjects receiving at least one dose of the investigational product.
Measure: Number; unit: episodes
Arm/Group | BID + Met | BID + Sita + Met | OD + Sita + Met
Number analyzed (Participants) | 192 | 193 | 190
episodes
  Diurnal (ADA) | 515 | 440 | 249
  Nocturnal (ADA) | 68 | 54 | 63
  Diurnal (additional minor) | 163 | 112 | 71
  Nocturnal (additional minor) | 21 | 14 | 23

11. Secondary Outcome: Change From Baseline in Patient Reported Outcome by Use of the Treatment Related Impact Measure - Diabetes.
Description: Estimated mean change from baseline in Treatment Related Impact Measure - Diabetes (TRIM-D) 'total score' to end of trial. The score measured treatment satisfaction. The scores were transformed to a 0-100 scale with higher scores indicating greater satisfaction.
Time Frame: Week 0 to Week 24
Population: Full analysis set (FAS) included all randomised subjects and missing data were imputed using last observation carried forward (LOCF). 545 subjects contributed to the statistical analysis at Week 24.
Measure: Least Squares Mean (Standard Error); unit: scores
Arm/Group | BID + Met | BID + Sita + Met | OD + Sita + Met
Number analyzed (Participants) | 178 | 184 | 183
scores | 6.22 (0.82) | 5.93 (0.81) | 6.20 (0.81)
Statistical Analysis 1: Comparison: BID + Met vs BID + Sita + Met; Test type: Superiority or Other; p = 0.800, Regression, Linear; Estimated treatment difference = 0.29, 95% CI [-1.97 to 2.56]
Statistical Analysis 2: Comparison: BID + Met vs OD + Sita + Met; Test type: Superiority or Other; p = 0.989, Regression, Linear; Estimated treatment difference = 0.02, 95% CI [-2.26 to 2.29]
Statistical Analysis 3: Comparison: BID + Sita + Met vs OD + Sita + Met; Test type: Superiority or Other; p = 0.809, Regression, Linear; Estimated treatment difference = -0.28, 95% CI [-2.52 to 1.97]

ADVERSE EVENTS:
Time Frame: Adverse events were captured the onset date on or after the first day of exposure to randomised treatment and no later than the last day of randomised treatment.
Description: Safety analysis set included all subjects receiving at least one dose of the investigational product.
Arm/Group | BID + Met | BID + Sita + Met | OD + Sita + Met
Serious Adverse Events (participants affected / at risk) | 7/192 | 5/193 | 4/190
Other Adverse Events (participants affected / at risk) | 30/192 | 25/193 | 32/190
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BID + Met (N=192) | BID + Sita + Met (N=193) | OD + Sita + Met (N=190)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Liver abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Burns second degree (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (4)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Thyroid cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoglycaemic unconsciousness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
VIIth nerve paralysis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BID + Met (N=192) | BID + Sita + Met (N=193) | OD + Sita + Met (N=190)
Diarrhoea (Gastrointestinal disorders) | 8 (10) | 1 (1) | 10 (10)
Influenza (Infections and infestations) | 11 (14) | 5 (6) | 10 (12)
Nasopharyngitis (Infections and infestations) | 9 (9) | 11 (12) | 8 (9)
Headache (Nervous system disorders) | 7 (11) | 11 (19) | 8 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Novo Nordisk maintains the right to be informed of any Investigator plans for publication and to review any scientific paper, presentation, communication or other information concerning the investigation described in this protocol. Novo Nordisk reserves the right to prior review of such publications and to ask for delay of publication of individual site results until after the primary manuscript is accepted for publication.